CLINICAL TRIAL: NCT03608722
Title: BrainCheck: Using Simple Video Games to Detect and Track Cognitive Health and Impairment
Brief Title: Video Games to Track Cognitive Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: BrainCheck, Inc. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1MAY15-93
Record Dates: First submitted 2018-05-22; First posted 2018-08-01 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Dementia; Mild Cognitive Impairment; Cognitive Impairment; Cognitive Decline; Cognitive Changes; Acute Changes in Cognition; Acute Head Injury; Concussion; Mild Traumatic Brain Injury
MeSH Terms: conditions — Dementia; Cognitive Dysfunction; Brain Concussion | interventions — Poverty Areas; Mental Status and Dementia Tests

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BrainCheck vs Pen and paper tests (Experimental): Compare patient performance on BrainCheck neurocognitive test vs pen and paper dementia tests (SLUMS, MMSE, MoCA), as well as an exploratory analysis comparing BrainCheck performance to aid in identifying patients with MCI and dementia vs physician diagnosis
  Interventions: Other: SLUMS; Other: MMSE; Other: MoCA; Device: BrainCheck
- BrainCheck performance in ESRD patients (Experimental): Assess BrainCheck test performance in patients with ESRD and how undergoing hemodialysis treatment can impact cognitive performance.
  Interventions: Device: BrainCheck

INTERVENTIONS:
Other: SLUMS — A pen and paper screening tool of cognitive impairment
  Other Names: St. Louis University Mental Status Exam
  Arms: BrainCheck vs Pen and paper tests
Other: MMSE — A pen and paper screening tool of cognitive impairment
  Other Names: The Mini-Mental State Examination or Folstein test
  Arms: BrainCheck vs Pen and paper tests
Other: MoCA — A pen and paper screening tool for cognitive impairment
  Other Names: Montreal Cognitive assessment
  Arms: BrainCheck vs Pen and paper tests
Device: BrainCheck — A computerized neurocognitive test administered via an electronic device, such as a phone, tablet or computer, that contains several assessments that will aid in establishing an individuals cognitive performance

SUMMARY:
The purpose of this study is to assess cognitive function using a rapid, portable, computerized neurocognitive testing device in a wide variety of clinical settings.

DETAILED DESCRIPTION:
Investigators will recruit participants from public places using the convenience sampling method. Informed consent will be obtain from all participants/parents as well as assent from minors. Participants will be asked to complete a brief yes/no questionnaire before the study begins. Participants will be asked to complete a 10 minute battery of tests consisting of simple video games designed to measure cognitive health. No personally identifiable information will be collected during the tests and all test data will remain anonymous. Data will be stored on servers with HIPAA-level security. No participants will be asked to modify their normal behavior in any way. No feedback or results will be given to participants. The tests will not be distressing in any way. To meet the objective of detecting cognitive impairment, investigators will test a broad array of participants from ages 10 through 99 in several different settings in parallel. The targeted cognitive stressors of advanced age, head injuries, physical strain, sleep deprivation, alcohol ingestion, and marijuana ingestion will be compared to healthy baseline controls. Collectively, these experiments aim to yield an end- deliverable of a rapid, non-invasive, portable piece of software that can be used to detect cognitive impairment.

A subset of participants will be asked to take the tests up to three times, so the total testing time is a max of 30 minutes. A subset of participants will be asked simple auxiliary questions, such as "Estimated in minutes, how long was your exercise or workout?". A subset of participants will be asked to wear a FitBit device to monitor their heart rate. A subset of participants will be asked to take a breathalyzer test (BACtrack S80).

ELIGIBILITY:
Inclusion Criteria:

* Aged 10 or older
* Function of both hands

Exclusion Criteria:

* Inability to speak English or Spanish
* Inability to read English or Spanish
* Unable to provide informed consent

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2500 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Identification of cognitive function performance utilizing a BrainCheck score | Throughout study completion, expected to be 3 years
  Utilizing BrainCheck to assess the ability of an individual to perform various mental activities on a score ranging from 0 to 30

SECONDARY OUTCOMES:
Identification of cognitive function performance on BrainCheck compared to pen and paper tests | Expect 2 years for subject enrollment. Data analysis to be completed 6 months after last subject enrolled
  Comparing BrainCheck's performance vs pen and paper dementia tests to establish sensitivity and specificity of BrainCheck to help identify patients with MCI and dementia

REFERENCES:
- [Derived] Groppell S, Soto-Ruiz KM, Flores B, Dawkins W, Smith I, Eagleman DM, Katz Y. A Rapid, Mobile Neurocognitive Screening Test to Aid in Identifying Cognitive Impairment and Dementia (BrainCheck): Cohort Study. JMIR Aging. 2019 Mar 21;2(1):e12615. doi: 10.2196/12615. PMID 31518280